CLINICAL TRIAL: NCT05725707
Title: Peer Led Friendship Group Intervention Development for Adults With Disabilities in Cambodia
Brief Title: Friendship Group Intervention Development in Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: University College Dublin (Other); Exceed Worldwide (Unknown)
Responsible Party: Principal Investigator, Dr Paul Best, Director, Queen's University, Belfast
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 028_2021
Record Dates: First submitted 2023-01-24; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Mental Health; Distress, Emotional; Worry
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Two groups -
  1. Group 1 - received a face-to-face based peer-led intervention
  2. Group 2 - received an online based peer-led intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face to face Friendship Group (Active Comparator): 8-week face-to-face peer-led intervention to support their mental health
  Interventions: Behavioral: Friendship Group
- Online Friendship Group (Active Comparator): 8 week online peer-led intervention to support their mental health
  Interventions: Behavioral: Friendship Group

INTERVENTIONS:
Behavioral: Friendship Group — Whether face-to-face or online delivery, each FG session followed the same broad format - (1) Group meditative exercise and reminder of group agreement (10 mins); (2) Check in with support group members and main session (50mins); (3) Summary of group discussion and homework activity planning (10mins); (4) Final group meditative exercise and closing of group (10mins). Session length was up to 80 minutes (see table 2) and each facilitator was provided with a manual describing each section as well as some hints and tips to promote discussion and engagement. While all FG's would follow this structure, group members would drive the content (particularly during Step 2).

SUMMARY:
A Friendship Group (FG's) (n= 4) will be delivered over an 8-week period (December 2021 - January 2022) to individuals who met the clinical distress threshold as per Kessler-10 score. FG's were offered face-to-face in Phnom Penh (n= 2) and online via Zoom (n= 2). Trained, community support workers and Prosthetists' from the Cambodian School of Prosthetics and Orthotics delivered FG's each week.

DETAILED DESCRIPTION:
Using a mixed methods design, the research team developed and implemented an 8-week peer-led intervention (known as a Friendship Group (FG) for Cambodian adults with physical disabilities using both face-to-face and online delivery methods.

Weekly Friendship Groups (n= 4) will be delivered over an 8-week period (December 2021 - January 2022) to individuals who met the clinical threshold as per Kessler-10 score (further details published elsewhere - blinded for review). FG's were offered face-to-face in Phnom Penh (n= 2) and online via Zoom (n= 2). Trained, community support workers and Prosthetists' from the Cambodian School of Prosthetics and Orthotics delivered FG's each week and followed the same four part structure described below. Prior to the first online session, each individual was asked to take part in a one-to-one orientation session to the platform to ensure that they could access the system without any issues. Participants were also reimbursed with costs for attending FG's (e.g. taxi fares for face-to-face or internet data for online groups). All those who had consented to receive communications were sent a weekly text message reminder 24 hours prior to the next FG meeting. All sessions were delivered in the local language (Khmer).

All participants in the study completed a screening survey to determine suitability. This included some basic socio-demographic information as well a series of validated psychometric scales described elsewhere.

Statistical Analysis

The data were screened for missing values and any error cases, such as extreme outliers. There were no missing values or error cases on any of the outcomes. The Wilcoxon Signed-Rank test was used to assess changes in pre-post scores for psychological distress, PTSD, worry, rumination and facets of mindfulness. With relatively small group sample sizes, differences between group allocations could confound intervention outcome measurement and it is therefore important in such circumstances to compare baseline differences between groups during the analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients and prospective patients attending Cambodian School of Prosthetics and Orthotics
* Meet the clinical threshold during Stage 1 screening
* Adults over the age of 18

Exclusion Criteria:

* Actively suicidal
* In receipt of additional specialist psychological therapy
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Kessler-10 | 8 weeks
  The primary outcome measure was Kessler-10 which is well suited to the Cambodian context and has been translated into Khmer and validated (38). Kessler-10 measures psychological distress and scoring ranges are as follows - likely to be well (score < 20), likely to have a mild distress (score = 20-24), likely to have moderate distress (score = 25-29) and likely to have a severe distress (score ≥ 30)

SECONDARY OUTCOMES:
Primary Care Screen | 8 weeks
  The Primary Care Screen is a five-item clinician administered screen that identifies individuals with probable PTSD. It has been used widely in primary care settings and begins by asking the individual whether they have been involved in any potentially traumatic event. Validation studies have demonstrated that answering 'yes' to three out of five questions is optimally sensitive to probable PTSD.
Pathological Worry | 8-weeks
  Pathological Worry: The 3-item Penn State Worry Questionnaire The 3-item Penn State Worry Questionnaire issued to measure pathological worry. The scale has comparable internal consistency and validity to the longer 16-item. Scores range from 5 (min) to 15 (max).

CONTACTS AND LOCATIONS:
Locations (1):
- Exceed Worldwide (DPO), Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No